CLINICAL TRIAL: NCT06050746
Title: Predictive Value of the PBS-score - A Prospective Observational Cohort Study Evaluating Recurrence of Idiopathic Clubfoot and Need for Additional Treatment
Brief Title: Predictive Value of the PBS-score in Children With Clubfoot
Status: Active, not recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Weidenhielm-Brostrom, Professor, Region Stockholm
Other Study IDs: k2022-10476-01
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Clubfoot
Keywords: PBS-score; Oxford Foot and Ankle Questionaire-child; Roye's score; Pedobarography
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Systematic screening — Included children will be followed prospectively during five years through clinical visits and medical records, where need for additional treatment (casting, braces and/or surgery) is the primary endpoint.
  Other Names: PBS-score, video evaluation, PROM, dynamic foot pressure

SUMMARY:
Evaluate the predictive value of the PBS-score in predicting recurrence of idiopathic clubfoot, measured as need for additional treatment.

DETAILED DESCRIPTION:
Using a consecutive inclusion, we aim to include 60 children and register data proposed by the COS for PEVA. All items of the PBS-score are video-documented, and dynamic foot pressure during walking is recorded during a clinical visit at the Motion Analysis Lab at Karolinska University Hospital. Children and caregivers will complete Roye's score, a disease-specific PROM and Oxford Foot and Ankle Questionaire-child (OxFAQc). For children aged 6 years or older, standing radiographic imaging of both feet will be performed. Inclusion criteria include: age 4-8 years, a diagnosis of idiopathic clubfoot, ability to walk 10 m repeatedly, and ability to communicate verbally (and in writing for caregivers) in Swedish or English. Included children will be followed prospectively during five years through clinical visits and medical records, where need for additional treatment (casting, braces and/or surgery) is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* age 4-10 years, a diagnosis of idiopathic clubfoot, ability to walk 10 m repeatedly, and ability to communicate verbally (and in writing for caregivers) in Swedish or English.

Exclusion Criteria:

* Syndromic clubfoot

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with idopatic clubfoot treated at Astrdi lindgren Children´s Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Need for further treatment | 5 years
  total number of casting, type of braces and/or choice of orthopedic surgery

SECONDARY OUTCOMES:
Patient reported outcome measures (PROM) | 5 years
  Children and caregivers will complete Roye's score, a disease-specific PROM. The Roye´s score consists of 10 items designed to measure treatment outcomes regarding overall satisfaction, appearance, pain, and physical limitations.
Patient reported outcome measures - The Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) is a child - or parent (proxy) | 5 years
  Children and caregivers will complete The Oxford Foot and Ankle Questionaire-child (OxFAQc) and a proxy for caregivers measure subjective well-being in children affected by foot and ankle pain and function. The OxFAQc has 15 items. The response options to each item are on a 5-point scale rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), where the number in brackets represents the value that should be applied by the scorer to each response. Domain scores are calculated as the total of the scale item scores divided by the maximum for each domain, physical 24, and school & play and emotional 16). Domain scores can be transformed to a percentage scale (0-100) to aid interpretation. A higher score for a domain represents better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Eva W Broström, Professor, Principal Investigator — Astrid Lindgren Children´s Hospital
Locations (1):
- Astrid Lindgren Children´s Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No